CLINICAL TRIAL: NCT03638453
Title: Pilot Feasibility of the Pediatric Cancer Resource Equity (PediCARE) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Charles H. Hood Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kira Bona, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-294; 1K07CA211847-01 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Other Cancer
Keywords: Pedi Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PediCARE (Experimental): * PediCARE Administered x6 mos
  * Resource Provision: Monthly Groceries (delivery via Instacart)
  * Resource Provision: Transport to/from home/hospital 8x per month (via RideHealth)
  Interventions: Other: PediCARE
- Usual Care (Active Comparator): The control group will receive usual supportive care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: PediCARE — PediCARE provides support for groceries (using an online grocery delivery service called Instacart) and transportation to and from the hospital (using rides through RideHealth).
  Arms: PediCARE
Other: Usual Care — Standard care per hospital guidelines.
  Arms: Usual Care

SUMMARY:
The goal of this new intervention is to make it easier for families to meet their basic household needs during childhood cancer treatment. The investigators want to learn how to best use PediCARE to help care for families.

DETAILED DESCRIPTION:
The investigators know from previous studies that in addition to the basic worries about a child's cancer therapy, many families experience financial stress during their child's treatment. Financial stress may include difficulty paying the rent or mortgage, keeping the electricity or heat on, or putting food on the table. One of the investigators' research goals is to find ways to decrease the financial impact of treatment on each family, and make sure that financial stress does not impact a child's experience during treatment.

The investigators have developed a new supportive care intervention called PediCARE (which stands for Pediatric Cancer Resource Equity) which provides support for groceries (using an online grocery delivery service called Instacart) and transportation to and from the hospital (using rides through services such as Uber and Lyft). The investigators have evaluated the PediCARE support program in a small group of parents and used feedback from these parents to improve PediCARE. The investigators are now ready to do a feasibility study to find out whether the investigators can reliably deliver the PediCARE intervention to families.

This type of study is called a feasibility study. The goal of this research study is to learn whether the investigators can successfully give the PediCARE support program to families-in other words, whether most families are interested in participating in a randomized study about the PediCARE support program and whether they use the PediCARE support program during the study. The investigators will also begin to understand whether the PediCARE support program reduces financial stress for families during therapy. Long-term, the investigators plan to test the PediCARE support program in a larger group of randomized families to answer the question of whether PediCARE reduces financial stress for families and improves outcomes during cancer treatment

ELIGIBILITY:
Inclusion Criteria:

* Child newly diagnosed with cancer within 2 months;
* Planned receipt of at least 4 cycles of chemotherapy at DFCI or UAB;
* Parent/guardian screened positive for HMH*;
* Child is <18 years at time of enrollment
* In accordance with previous research1 families will be operationalized as having HMH for eligibility purposes if they report at least one of the below four concrete needs assessed during routine clinical care as follows:

  * Food insecurity.
  * Housing Insecurity.
  * Energy Insecurity.
  * Transportation Insecurity.

HMH screening is performed as standard of care by site-specific psychosocial providers.

Exclusion Criteria:

* Child with diagnosis of relapsed cancer;
* Child planned to receive fewer than 4 cycles of chemotherapy
* Child planned to receive observation, radiation or surgical resection only;
* Planned transfer of child to a non-DFCI or UAB facility for chemotherapy treatment;
* Foreign national family receiving cancer care as an Embassy-pay patient;
* Child is enrolled on DFCI 16-001 (due to ongoing embedded descriptive HMH study)

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kira Bona, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newman H, Jones E, Li Y, Umaretiya PJ, Wolfson JA, Wolfe J, Bona K. Providing Groceries and Transportation to Poverty-Exposed Pediatric Oncology Families: The PediCARE Pilot Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2412890. doi: 10.1001/jamanetworkopen.2024.12890. PMID 38819828

RESULTS

PARTICIPANT FLOW:
Groups:
- PediCARE: * PediCARE Administered x6 mos
  * Resource Provision: Monthly Groceries (delivery via Instacart)
  * Resource Provision: Transport to/from home/hospital 8x per month (via RideHealth)
  PediCARE: PediCARE provides support for groceries (using an online grocery delivery service called Instacart) and transportation to and from the hospital (using rides through RideHealth).
Period: Overall Study
Arm/Group | PediCARE | Usual Care
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PediCARE | Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (6.3) | 8.3 (5.8) | 8.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 8 | 9 | 17
  White | 10 | 10 | 20
  Missing | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Recruited
Description: At least 75 percent consent to randomization (e.g. recruitment).
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | PediCARE | Usual Care
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

2. Primary Outcome: Percentage of Attrition
Description: At most 20 percent attrition per arm.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | PediCARE | Usual Care
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

3. Secondary Outcome: Change in Household Material Hardship (HMH) in PediCARE vs Usual Care
Description: Change in HMH score (0-4) at intervention completion (6-months) compared to baseline. For each family, the difference between 6-month and baseline HMH scores will be categorized as 1) stabilized or decreased or 2) increased HMH exposure. For each arm, the proportion of families with stabilized or decreased HMH at the completion of the intervention (6-months) will be estimated.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | PediCARE | Usual Care
Number analyzed (Participants) | 20 | 20
Participants | 17 | 14

4. Secondary Outcome: Proportion of Patients With at Least One Emergency Department (ED) Visit or Intensive Care Unit (ICU) for Each Arm
Description: The proportion of patients with at least one ED and/or ICU visit will be estimated for PediCARE and Usual Care groups.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | PediCARE | Usual Care
Number analyzed (Participants) | 20 | 20
Participants | 13 | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the study period of 6 months.
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information does not differ from the clinicaltrials.gov definitions.
Arm/Group | PediCARE | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
At study conclusion, investigators identified concerns regarding the validity of ED visits given reported frequency of participants potentially being seen at ED's outside of the enrolling site that could not be quantified via chart abstraction. As a result, it was determined that data analysis for effect size estimation using this endpoint would not be informative from this pilot study, and these data were not reported in the primary manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT03638453/Prot_SAP_000.pdf